CLINICAL TRIAL: NCT03601715
Title: Coplanar Arrangement of Shortwave Diathermy is the Most Efficient in Skin Temperature Change: A Randomized Crossover Trial
Brief Title: Analysis of Human Tissue Temperature After Application of Therapeutic Modalities.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alessandro Haupenthal (Other)
Collaborators: Santa Catarina Federal University (Other)
Responsible Party: Sponsor-Investigator, Alessandro Haupenthal, Principal Investigator, Universidade Federal de Santa Catarina
Organization: Universidade Federal de Santa Catarina (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1.771.454
Record Dates: First submitted 2018-07-03; First posted 2018-07-26 (Actual); Results first posted 2020-01-02 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Humans; Young Adult; Health
Keywords: Diathermy; Short-Wave Therapy; Body temperature; Skin Temperature
MeSH Terms: conditions — Fever

STUDY DESIGN:
Intervention Model Description: A randomized single blind, crossover experimental study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Coplanar (Active Comparator): Electrode placed side by side on the same aspect of the right tight.
  Interventions: Other: Coplanar
- Contraplanar (Active Comparator): Electrode placed over opposite aspects of the right tight.
  Interventions: Other: Contraplanar
- Longitudinal (Active Comparator): One electrode is placed at each end of the limb in opposite aspects of the tight.
  Interventions: Other: Longitudinal

INTERVENTIONS:
Other: Coplanar — The coplanar arrangement will be applicated in each one of the subjects. The intervention will last 20 minutes. A towel will be placed between the pad electrode and the skin to improve contact, besides, the tight and the electrode will be wrapped with an elastic band for the same purpose. The subject will receive orientation related to the heat intensity, it must be a comfortable perception of heat (the intensity will be regulated on the equipment to guarantee that).
  Arms: Coplanar
Other: Contraplanar — The contraplanar arrangement will be applicated in each one of the subjects. The intervention will last 20 minutes. A towel will be placed between the pad electrode and the skin to improve contact, besides, the tight and the electrode will be wrapped with an elastic band for the same purpose. The subject will receive orientation related to the heat intensity, it must be a comfortable perception of heat (the intensity will be regulated on the equipment to guarantee that).
  Arms: Contraplanar
Other: Longitudinal — The longitudinal arrangement will be applicated in each one of the subjects. The intervention will last 20 minutes. A towel will be placed between the pad electrode and the skin to improve contact, besides, the tight and the electrode will be wrapped with an elastic band for the same purpose. The subject will receive orientation related to the heat intensity, it must be a comfortable perception of heat (the intensity will be regulated on the equipment to guarantee that).
  Arms: Longitudinal

SUMMARY:
Attempting an effective treatment is essential to the physiotherapist to understand how his conducts affect body tissues and the whole system, besides understand properly how and when therapeutic modalities could be use in the rehabilitation process. There are several research articles pointing the use of heat as an efficient agent to accelerate tissue healing. Clarifying the remaining doubts related to therapeutic modalities use can be beneficial for functional rehabilitation.

In physiotherapy, shortwave diathermy is one of the standards treatments for heat inducement. The capacitance shortwave technique consists in the use of two pad electrodes that can be positioned in three different arrangements: coplanar (placed side by side on the same aspect of the part to be treated), contraplanar (placed over opposite aspects of the body part to be treated) and longitudinal (one electrode is placed at each end of the limb in opposite aspects of the body par to be treated). There is no evidence of which arrangement is the most efficient.

Besides shortwave diathermy being a very established therapeutic modality, the use of this recourse in the most effective way rely on the properly answer of the remaining questions related to its application. Therefore, the purpose of this study is to analyze which one of the capacitance shortwave technique is the most efficient in inducing and maintaining heat.

Given the high-frequency waves field orientation could be suggested that the coplanar arrangement will lead to bigger heat inducement, and will maintain it for longer time.

DETAILED DESCRIPTION:
The data for the sample size calculation was taken from a pilot study of 8 subjects. The software used to calculate the sample was GPower 3.1.9.2. A 18 subjects sample were obtained to reach a power of 90%, needed to detect a difference on the average of the groups in repeated measures with an alpha of 5%. The sample size was raised to 20 subjects for eventually lost. The subjects will be chosen through social media and informal invitations.

The subjects will attend to the laboratory four times, the first day for orientation and measurements (body mass and skinfold), the data collection will start on the second day.

The room temperature will be set between 23 °C and 25 °C, and the humidity around 70%. The subject will be placed in supine position on the stretcher, instructed to relax and not touch the right thigh region for 20 minutes before the intervention (for body temperature stabilization).

The thigh size will be measured form the base of the patella to the anterior superior iliac spine and the center marked to determine the place where the temperature will be collected. The minimum space between electrodes position will be at least of the size of one electrode. The temperature of the right thigh will be measured by infrared thermography before the intervention, right after the removal and every minute until the total time of the intervention.

To summarize the data, it will be used descriptive statistics, the values of average, standard deviation and the collected measurements will be identified. Through Shapiro-Wilk test the distribution of data regarding normality will be verified. To compare the initial and the final test values the ANOVA and the post-hoc of Bonferroni will be used. In the case of data being out of the normal standards, a transformation will be used to reach the normality. If the data still don't reach the normality after the transformation, the non-parametric tests will be used (Mann-Whitney e Kruskal Walis). The confidence level adopted for all tests will be 95% (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* No orthopedic injury in three months prior to the study;
* A minimum of 19 years of age, and a maximum of 40 years;
* Male;
* Must agree not to practice exercise the day before the study and not ingest caffeine, alcohol, or food one hour before intervention.

Exclusion Criteria:

* Skinfold minor than 2cm;
* Circulatory system disease;
* Ischemic tissue or malignant tumors;
* External fixation, metal or pacemaker;
* Any thigh open wound;
* Muscular or neurological disease;
* Diabetes diagnosed;
* Cigarette smoker.

Ages: 19 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Haupenthal, Doctorate, Study Director — Santa Catarina Federal University
Locations (1):
- Santa Catarina Federal University, Araranguá, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Means and standard deviations of temperature change.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Background] ABIB, R. T. et al. Avaliação da diatermia por ondas curtas contínuo na temperatura superficial do músculo quadríceps. Ciência em Movimento, v. 1, n. 23, p. 69-77, 2010.
- [Background] BRASILEIRO, J. S.; FARIA, A. F.; QUEIROZ, L. L. Influància do resfriamento e do aquecimento local na flexibilidade dos músculos isquiotibiais. Revista Brasileira de Fisioterapia, v. 11, n. 1, p. 57-61, 2007.
- [Background] Delpizzo V, Joyner KH. On the safe use of microwave and shortwave diathermy units. Aust J Physiother. 1987;33(3):152-62. doi: 10.1016/S0004-9514(14)60592-4. PMID 25025704
- [Background] Draper DO, Knight K, Fujiwara T, Castel JC. Temperature change in human muscle during and after pulsed short-wave diathermy. J Orthop Sports Phys Ther. 1999 Jan;29(1):13-8; discussion 19-22. doi: 10.2519/jospt.1999.29.1.13. PMID 10100117
- [Background] Draper DO, Miner L, Knight KL, Ricard MD. The Carry-Over Effects of Diathermy and Stretching in Developing Hamstring Flexibility. J Athl Train. 2002 Mar;37(1):37-42. PMID 12937442
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Garrett CL, Draper DO, Knight KL. Heat distribution in the lower leg from pulsed short-wave diathermy and ultrasound treatments. J Athl Train. 2000 Jan;35(1):50-5. PMID 16558608
- [Background] Hawkes AR, Draper DO, Johnson AW, Diede MT, Rigby JH. Heating capacity of rebound shortwave diathermy and moist hot packs at superficial depths. J Athl Train. 2013 Jul-Aug;48(4):471-6. doi: 10.4085/1062-6050-48.3.04. Epub 2013 Mar 19. PMID 23855362
- [Background] Ichinoseki-Sekine N, Naito H, Saga N, Ogura Y, Shiraishi M, Giombini A, Giovannini V, Katamoto S. Changes in muscle temperature induced by 434 MHz microwave hyperthermia. Br J Sports Med. 2007 Jul;41(7):425-9. doi: 10.1136/bjsm.2006.032540. Epub 2007 Jan 29. PMID 17261552
- [Background] Peres SE, Draper DO, Knight KL, Ricard MD. Pulsed Shortwave Diathermy and Prolonged Long-Duration Stretching Increase Dorsiflexion Range of Motion More Than Identical Stretching Without Diathermy. J Athl Train. 2002 Mar;37(1):43-50. PMID 12937443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Paticipants, reached through social media, volunteered to participate in the study.Participant enrollment began on 9/3/18 and the last participant was enrolled on 11/9/18.
Pre-assignment Details: All the twenty health enrolled male subjects met the inclusion criteria and were randomly allocated an order in which treatments were received.
Groups:
- Coplanar First, Then Contraplanar and at Last Longitudinal: After 20 minutes of acclimatization, participants received the capacitive arrangement as determined for 20 minutes. First, received Coplanar arrangement application, then, after a washout period of at least one day received Contraplanar application and after a washout period of at least one day received Longitudinal application.
- Contraplanar First, Then Coplanar and at Last Longitudinal: After 20 minutes of acclimatization, participants received the capacitive arrangement as determined for 20 minutes. First, received Contraplanar arrangement application, then, after a washout period of at least one day received Coplanar application and after a washout period of at least one day received Longitudinal application.
- Longitudinal First, Then Coplanar and at Last Contraplanar: After 20 minutes of acclimatization, participants received the capacitive arrangement as determined for 20 minutes. First, received Longitudinal arrangement application, then, after a washout period of at least one day received Coplanar application and after a washout period of at least one day received Contraplanar application.
Period: First Intervention
Arm/Group | Coplanar First, Then Contraplanar and at Last Longitudinal | Contraplanar First, Then Coplanar and at Last Longitudinal | Longitudinal First, Then Coplanar and at Last Contraplanar
Started | 7 | 7 | 6
Completed | 7 | 7 | 6
Not Completed | 0 | 0 | 0
Period: Washout 1 (at Least 24 Hours)
Arm/Group | Coplanar First, Then Contraplanar and at Last Longitudinal | Contraplanar First, Then Coplanar and at Last Longitudinal | Longitudinal First, Then Coplanar and at Last Contraplanar
Started | 7 | 7 | 6
Completed | 7 | 7 | 6
Not Completed | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Coplanar First, Then Contraplanar and at Last Longitudinal | Contraplanar First, Then Coplanar and at Last Longitudinal | Longitudinal First, Then Coplanar and at Last Contraplanar
Started | 7 | 7 | 6
Completed | 6 | 6 | 6
Not Completed | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Period: Wash Out 2 (at Least 24 Hours)
Arm/Group | Coplanar First, Then Contraplanar and at Last Longitudinal | Contraplanar First, Then Coplanar and at Last Longitudinal | Longitudinal First, Then Coplanar and at Last Contraplanar
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Coplanar First, Then Contraplanar and at Last Longitudinal | Contraplanar First, Then Coplanar and at Last Longitudinal | Longitudinal First, Then Coplanar and at Last Contraplanar
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coplanar First, Then Contraplanar and at Last Longitudinal | Contraplanar First, Then Coplanar and at Last Longitudinal | Longitudinal First, Then Coplanar and at Last Contraplanar | Total
Number analyzed (Participants) | 7 | 7 | 6 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.7 (1.6) | 22.2 (1.79) | 20 (2.09) | 21.4 (2.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 7 | 7 | 6 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 7 | 7 | 6 | 20
Height [Mean (Standard Deviation); unit: meters] | 1.74 (0.08) | 1.75 (0.04) | 1.78 (0.08) | 1.76 (0.07)
Mass [Mean (Standard Deviation); unit: Kilograms] | 74 (12.02) | 73 (14.4) | 72.6 (6.63) | 73.2 (10.6)
Body mass index [Mean (Standard Deviation); unit: Kilograms/meters²] | 24.2 (3.09) | 23.4 (3.37) | 22.9 (2.2) | 23.6 (2.46)

OUTCOME MEASURES:

1. Primary Outcome: The Most Effective Capacitance Shortwave Technique in Relation to Temperature Increase and Heat Conservation Measured by Infrared Thermography
Description: Evaluation of the most effective electrode arrangement (coplanar, contraplanar or longitudinal) in relation to temperature increase and heat conservation. Measured using a infrared camera in three sessions, with a washout period of at least 24 hours.
Time Frame: 3 days
Population: Occurred 2 losses to follow up.
Measure: Mean (Standard Deviation); unit: Celsius
Groups:
- Coplanar: Electrode placed as far apart as the cross-sectional diameter of the pad electrode on the same aspect of the right tight.
  After 20 minutes of acclimatization, participants received application for 20 minutes. The electrode pads were surrounded by felt and positioned over 1 cm of toweling, besides, we wrapped the tight and the electrodes using an elastic band. We controlled the intensity based on a referred warm heat perception by the subject.
- Contraplanar: Electrode placed over opposite aspects in the right tight centre.
  After 20 minutes of acclimatization, participants received application for 20 minutes. The electrode pads were surrounded by felt and positioned over 1 cm of toweling, besides, we wrapped the tight and the electrodes using an elastic band. We controlled the intensity based on a referred warm heat perception by the subject.
- Longitudinal: Each electrode is placed at the final portion of the limb in opposite aspects of the right tight.
  After 20 minutes of acclimatization, participants received application for 20 minutes. The electrode pads were surrounded by felt and positioned over 1 cm of toweling, besides, we wrapped the tight and the electrodes using an elastic band. We controlled the intensity based on a referred warm heat perception by the subject.
Arm/Group | Coplanar | Contraplanar | Longitudinal
Number analyzed (Participants) | 18 | 18 | 18
Celsius
  Thigh centre (after electrodes removal) | 1.72 (1.01) | 0.58 (0.99) | 0.94 (0.51)
  Under the electrode (after electrodes removal) | 7.9 (1.76) | 6.52 (2.68) | 7.46 (1.8)
  Thigh centre (5 min after removal) | 1.33 (0.9) | 0.12 (0.9) | 0.61 (0.44)
  Under the electrode (5 min after removal) | 2.76 (1.17) | 2.35 (1.53) | 2.65 (1.3)
  Thigh centre (10 min after removal) | 1.17 (1.01) | -0.06 (0.98) | 0.45 (0.55)
  Under the electrode (10 min after removal) | 2.15 (1.21) | 1.87 (1.36) | 2.06 (1.1)
  Thigh centre (15 min after removal) | 1.07 (1.06) | -0.17 (1.02) | 0.32 (0.69)
  Under the electrode (15 min after removal) | 1.8 (1.22) | 1.48 (1.29) | 1.74 (1.07)
  Thigh centre (20 min after removal) | 0.83 (1.19) | -0.07 (1.06) | 0.22 (0.78)
  Under the electrode (20 min after removal) | 1.41 (1.27) | 1.28 (1.28) | 1.43 (1.07)
  Thigh centre (25 min after removal) | 0.78 (1.17) | -0.09 (1.09) | 0.16 (0.73)
  Under the electrode (25 min after removal) | 1.14 (1.22) | 1.1 (1.16) | 0.94 (1.29)
Statistical Analysis 1: Comparison: Coplanar vs Contraplanar vs Longitudinal; Based on a pilot test with eight subjects, we calculated that we would need 18 subjects to give 90% power to detect the most efficient arrangement with a α level of .05. Considering losses to follow up , we increased the sample size by 10%; Test type: Superiority; p < 0.05, ANOVA — Bonferroni post-hoc tests; Effect size was calculated through partial eta squared and correlated using Cohen index (.1 to .3 as small, .3 to .5 as medium, and over .5 as large)

2. Secondary Outcome: Temperature Increase
Description: Determine which capacitance shortwave technique will increase the temperature the most after 20 minutes of application. The skin temperature will be verified by infrared thermography. This evaluation will occur in three 24 hours apart visits, each for one of the three capacitance shortwave technique.
Time Frame: 3 days
Population: Occurred 2 losses to follow up.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Coplanar | Contraplanar | Longitudinal
Number analyzed (Participants) | 18 | 18 | 18
Celsius
  On thigh centre, after electrodes removal | 1.72 (1.01) | 0.58 (0.99) | 0.94 (0.51)
  Under the electrode (after electrodes removal) | 7.9 (1.76) | 6.52 (2.68) | 7.46 (1.8)
Statistical Analysis 1: Comparison: Coplanar vs Contraplanar vs Longitudinal; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, ANOVA — Bonferroni post-hoc tests; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Heat Conservation
Description: Determinate which capacitance shortwave technique retain the induced heat for longer time. The skin temperature will be verified by infrared thermography before the application and after during 25 minutes, 1 minutes apart each measure. This evaluation will occur in three 24 hours apart visits, each for one of the three capacitance shortwave technique.
Time Frame: 3 days
Population: Occurred 2 losses to follow up.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Coplanar | Contraplanar | Longitudinal
Number analyzed (Participants) | 18 | 18 | 18
Celsius
  Thigh centre (5 min after removal) | 1.33 (0.9) | 0.12 (0.9) | 0.61 (0.44)
  Under the electrode (5 min after removal) | 2.76 (1.17) | 2.35 (1.53) | 2.65 (1.3)
  Thigh centre (10 min after removal) | 1.17 (1.01) | -0.06 (0.98) | 0.45 (0.55)
  Under the electrode (10 min after removal) | 2.15 (1.21) | 1.87 (1.36) | 2.06 (1.1)
  Thigh centre (15 min after removal) | 1.07 (1.06) | -0.17 (1.02) | 0.32 (0.69)
  Under the electrode (15 min after removal) | 1.8 (1.22) | 1.48 (1.29) | 1.74 (1.07)
  Thigh centre (20 min after removal) | 0.83 (1.19) | -0.07 (1.06) | 0.22 (0.78)
  Under the electrode (20 min after removal) | 1.41 (1.27) | 1.28 (1.28) | 1.43 (1.07)
  Thigh centre (25 min after removal) | 0.78 (1.17) | -0.09 (1.09) | 0.16 (0.73)
  Under the electrode (25 min after removal) | 1.14 (1.22) | 1.1 (1.16) | 0.94 (1.29)
Statistical Analysis 1: Comparison: Coplanar vs Contraplanar vs Longitudinal; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, ANOVA — Bonferroni post-hoc tests; [other analysis details as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: The participants were monitored for adverse events over the duration of treatment (at least 5 days, considering the washout period minimum of 1 day).
Description: Other adverse events refers to burns.
Arm/Group | Coplanar | Contraplanar | Longitudinal
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT03601715/Prot_SAP_000.pdf